CLINICAL TRIAL: NCT00295139
Title: Behavioral Treatment of Drug Abuse in SPMI Patients
Brief Title: Behavioral Treatment of Drug Abuse in Severe and Persistent Mental Illness (SPMI) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Melanie Bennett, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00041195
Record Dates: First submitted 2006-02-19; First posted 2006-02-22 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia; Mood Disorders; Substance Dependence
Keywords: treatment; dual diagnosis
MeSH Terms: conditions — Schizophrenia; Mood Disorders; Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Behavioral Treatment for Substance Abuse in SPMI (BTSAS)
  Interventions: Behavioral: Behavioral Treatment for Substance Abuse in SPMI (BTSAS)
- 2 (Experimental): Behavioral Treatment for Substance Abuse in SPMI (BTSAS) + Critical Time Intervention (CTI)
  Interventions: Behavioral: Behavioral Treatment for Substance Abuse in SPMI (BTSAS); Behavioral: Critical Time Intervention (CTI)
- 3 (Active Comparator): Supportive Treatment in Addiction Recovery (STAR)
  Interventions: Behavioral: Supportive Treatment in Addiction Recovery (STAR)

INTERVENTIONS:
Behavioral: Behavioral Treatment for Substance Abuse in SPMI (BTSAS) — Multifaceted treatment for substance abuse in dual disordered patients which contains 6 components: 1) a urinalysis contingency to enhance motivation to change and increase the salience of goals; 2) structured goal setting to identify realistic, short term goals for decreased substance use; 3) motivational interviewing to enhance motivation to reduce use; 4) social skills and drug refusal skills to enable development of relationships with people who do not use drugs, and to provide success experiences that can increase self-efficacy for change; 5) education about the reasons for substance use and the particular dangers of substance use for people with SPMI; and 6) relapse prevention training that focuses on behavioral skills for coping with urges and dealing with high risk situations and lapses. BTSAS is specifically structured to reduce the load on memory and attention, and minimize demands on higher level cognitive processes.
  Arms: 1; 2
Behavioral: Supportive Treatment in Addiction Recovery (STAR) — Manualized substance abuse treatment as usual
  Arms: 3
Behavioral: Critical Time Intervention (CTI) — Case management component
  Arms: 2

SUMMARY:
The main purpose of this study is to determine if the multifaceted treatment for substance abuse in dual disordered patients is more effective in reducing drug use than a supportive control treatment. The researchers will also determine if adding a case management component (Critical Time Intervention; CTI) to the intervention will increase treatment engagement and retention.

DETAILED DESCRIPTION:
Drug and alcohol abuse by people with severe and persistent mental illness (SPMI) is one of the most significant problems facing the public mental health system. We have been conducting a project to develop a multifaceted treatment for substance abuse in dual disordered patients (Behavioral Treatment for Substance Abuse in Schizophrenia; BTSAS). Results have shown that the treatment is well-accepted by patients and has a significant effect on drug use. While BTSAS has been effective at retaining subjects and fostering reduced drug use, a major problem that occurred was low rates of engagement. The main purpose of this study is to determine if BTSAS is more effective in reducing drug use than a supportive control treatment and to determine if adding a case management component (Critical Time Intervention; CTI) will increase treatment engagement and retention in BTSAS.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of schizophrenia or schizoaffective disorder or a diagnosis of other severe mental disorder including bipolar disorder, major depression, or severe anxiety disorder (by definition, the patient has worked 25% or less of the past year; and/or the patient receives payment for mental disability)
* a diagnosis of current dependence for opiates, cocaine, or marijuana
* ability and willingness to attend treatment sessions for 6 months
* ability and willingness to provide consent to participate
* enrolled in mental health care

Exclusion Criteria:

* documented history of severe neurological disorder or severe head trauma with loss of consciousness
* severe or profound mental retardation as indicated by chart review
* inability to effectively participate in the baseline assessments due to intoxication or psychiatric symptoms on two successive appointments
* had a substantial trial in either intervention of the Evaluation of Behavioral Treatment for Substance Abuse in Schizophrenia protocol (H-20680)
* inability to attend group sessions due to transportation or other logistical problems
* inability to attend scheduled treatment sessions on a regular basis for any reason, or to appropriately participate in research activities due to behavioral or psychiatric problems

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 293 (Actual)
Dates: Start 2005-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Urinalysis | Baseline, 2 and 4 months, post and 6-month follow-up, and at each treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Bellack, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - Health Care for the Homeless, Baltimore, Maryland
  - University of Maryland, Baltimore, Baltimore, Maryland
  - VA Maryland Health Care System, Baltimore, Maryland
  - Mosaic Community Services, Catonsville, Maryland

REFERENCES:
- [Background] Bellack AS, Gearon JS. Substance abuse treatment for people with schizophrenia. Addict Behav. 1998 Nov-Dec;23(6):749-66. doi: 10.1016/s0306-4603(98)00066-5. PMID 9801714
- [Background] Bellack AS, DiClemente CC. Treating substance abuse among patients with schizophrenia. Psychiatr Serv. 1999 Jan;50(1):75-80. doi: 10.1176/ps.50.1.75. PMID 9890583
- [Background] Gearon JS, Bellack AS. Women with schizophrenia and co-occurring substance use disorders: an increased risk for violent victimization and HIV. Community Ment Health J. 1999 Oct;35(5):401-19. doi: 10.1023/a:1018778310859. PMID 10547116
- [Background] Bellack, A.S. (2000) Behavioral treatment for substance abuse in schizophrenia. The Addictions Newsletter, 7, 20-22
- [Background] Gearon JS, Bellack AS. Sex differences in illness presentation, course, and level of functioning in substance-abusing schizophrenia patients. Schizophr Res. 2000 May 25;43(1):65-70. doi: 10.1016/s0920-9964(99)00175-9. PMID 10828416
- [Background] Gearon JS, Bellack AS, Rachbeisel J, Dixon L. Drug-use behavior and correlates in people with schizophrenia. Addict Behav. 2001 Jan-Feb;26(1):51-61. doi: 10.1016/s0306-4603(00)00084-8. PMID 11196292
- [Background] Bennett ME, Bellack AS, Gearon JS. Treating substance abuse in schizophrenia. An initial report. J Subst Abuse Treat. 2001 Mar;20(2):163-75. doi: 10.1016/s0740-5472(00)00167-7. PMID 11306219
- [Background] Gearon JS, Kaltman SI, Brown C, Bellack AS. Traumatic life events and PTSD among women with substance use disorders and schizophrenia. Psychiatr Serv. 2003 Apr;54(4):523-8. doi: 10.1176/appi.ps.54.4.523. PMID 12663840
- [Background] Gearon JS, Nidecker M, Bellack A, Bennett M. Gender differences in drug use behavior in people with serious mental illnesses. Am J Addict. 2003 May-Jun;12(3):229-41. PMID 12851019
- [Background] Bellack AS, Bennett ME, Gearon JS, Brown CH, Yang Y. A randomized clinical trial of a new behavioral treatment for drug abuse in people with severe and persistent mental illness. Arch Gen Psychiatry. 2006 Apr;63(4):426-32. doi: 10.1001/archpsyc.63.4.426. PMID 16585472